CLINICAL TRIAL: NCT00102635
Title: A Phase IB Randomized Translational Study of Fenretinide (4-HPR) in Combination With SCH66336, a Farnesyl Transferase Inhibitor, in Patients With Advanced or Recurrent Head and Neck Cancer
Brief Title: 4-HPR and FTI in Head and Neck Squamous Cell Carcinoma (HNSCC)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Slow accrual.
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ID01-455; NCT00103090 (obsolete NCT alias)
Record Dates: First submitted 2005-01-31; First posted 2005-02-01 (Estimated); Last update posted 2018-11-15 (Actual); Status verified 2018-11

CONDITIONS: Head and Neck Cancer
Keywords: apoptotic activity; 4-HPR; FTI; Fenretinide; SCH66336; Farnesyl Transferase Inhibitor; HNC
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Fenretinide; lonafarnib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 4-HPR + FTI (Experimental): SCH66336 daily for 21 days each cycle and with 4-HPR daily on days 1-7 only. On day 1 of cycle 1, 4-HPR only beginning SCH66336 on day 2 of cycle 1.
  Interventions: Drug: Fenretinide (4-HPR); Drug: SCH66336

INTERVENTIONS:
Drug: Fenretinide (4-HPR) — Oral 100 mg capsules in two divided doses at least 8 hours apart for 7 days each cycle.
Drug: SCH66336 — Oral capsules with 50 mg, 75 mg, or 100 mg formulation in two divided doses at least 8 hours apart for 21 days each cycle.
  Other Names: Lonafarnib; SCH 66336; Sarasar

SUMMARY:
The primary objective of this study is to estimate the modulation of intermediate biological endpoints of the combination of 4-HPR and SCH66336, a farnesyl transferase inhibitor (FTI), across 4 randomly assigned dose levels in patients with locally advanced or recurrent head and neck cancer. We will also assess the activity, safety, tolerability and side effects of 4-HPR/SCH66336 and hope to establish a phase II regimen.

DETAILED DESCRIPTION:
The drug fenretinide is a retinoid that is similar to vitamin A. It is believed that fenretinide can cause cancer cells to die. SCH66336 is a drug that blocks farnesyl protein transferase (a substance needed by cancer cells to grow). It is believed that SCH66336 may selectively stop cancer cells from growing while not affecting normal cells.

Both SCH66336 and fenretinide are taken orally and must be swallowed whole (i.e., the drugs may not be broken to make swallowing easier). Individuals who cannot take the study medications whole by mouth cannot enroll in this study.

In this study participants will receive SCH66336 twice a day for each day of a 21-day cycle. Participants will also take fenretinide twice a day on Days 1-7 of the same cycle. Before beginning treatment, participants will have a complete physical exam, including measurement of height, weight, and vital signs. Participants will have blood and urine tests, a chest x-ray, and an ECG (heart function test). Females who are able to become pregnant must have a negative blood pregnancy test. In addition, all participants will have a neurological exam and will complete a questionnaire about their night vision. Some individuals may need an eye exam.

Before beginning treatment, participants will have a biopsy of their tumor and will provide a sample of their buccal mucosa (inner cheek). In the biopsy, a sample of tumor tissue will be removed with a large needle. The buccal mucosa sample will be obtained by scraping the inside of the cheek. Participants will also have an extra blood sample (about 2 tablespoons) drawn. The tumor, buccal mucosa, and blood samples are all being obtained for research purposes only and will not directly benefit the participant.

During the study, a physician will examine participants at least once a week for the first cycle of treatment. A treatment cycle is 3 weeks. Participants will also have weekly blood tests. After the first cycle of treatment, participants will have exams every 3 weeks. In addition, participants will have urine tests every 3 weeks, a neurological exam after the first 3 weeks and then as needed, and a chest x-ray every 3 weeks. Every 3 months, participants will complete a questionnaire about their night vision and will have an eye exam, if needed.

While on this study, individuals will also participate in a pharmacokinetic study to measure the levels of the drugs in the blood. On the first day of treatment, the participant will have blood samples (about 1 teaspoon each) drawn before taking fenretinide and then 1, 2, 4, 6, 9, and 12 hours after taking fenretinide. The participant will not take the first dose of SCH66336 until after these blood samples have been taken. Additional blood samples (about 1 teaspoon each) will be taken at these same times on Day 7 of the first treatment cycle and on Day 1 of the second treatment cycle. A single blood sample (about 1 teaspoon) will be taken before taking the study drugs on Day 7 of treatment Cycles 3, 4, 5, and 6.

Participants will have biopsies of their tumors, extra blood tests and will provide buccal mucosa samples on Days 7 and 21 of the first treatment cycle. These biopsies, cheek scrapings, and extra blood tests are for research purposes only and will not directly benefit the participant. Approximately two tablespoons of blood will be drawn during each of these extra blood tests. This blood, buccal mucosa (cheek), and tumor tissue will be studied to learn how the treatment drugs work in the body and what effects they have. Participants may remain on the study as long as they are responding to the SCH66336/fenretinide combination and as long as their physician feels it is of benefit.

After completing treatment, participants will be contacted about every 3 months to check on the disease status. Participants will come to M.D. Anderson for clinical evaluations every 3 months for a period of 24 months.

Fenretinide is in the form of capsules and SCH66336 is in the form of tablets. Participants will take the fenretinide capsules by mouth twice a day for seven days in a row at the start of each treatment cycle. Participants will take the SCH66336 tablets twice a day for 21 days in a row in each cycle. Participants will be given a "pill diary" in which they should record when they take the study medications and how many capsules and tablets they take. Participants will bring this diary and any unused medication when they return to the clinic for their check-ups. At the beginning of a treatment cycle, participants should take both drugs together at least 8 hours apart with either a high-fat meal or a glass of whole milk. Participants should continue taking the SCH66336 tablets at least 8 hours apart and with a meal or a glass of whole milk during Days 8-21 of each treatment cycle. Participants will not take fenretinide capsules during Days 8-21 of a treatment cycle.

While on this study, participants may not drink grapefruit juice.

This is an investigational study. The FDA has authorized the use of this drug combination in research but has not approved it for widespread use. About 40 individuals will take part in this study. All will be enrolled at M.D. Anderson Cancer Center.

ELIGIBILITY:
Inclusion Criteria:

* Patient has histologically proven squamous cell carcinoma of the head and neck which is biopsy accessible and is not considered curable by standard measures.
* Patient has a Karnofsky performance status >/= 70%
* Patient has adequate bone marrow function: *WBC >/= 3,000 cells/mm^3, *ANC >/= 1,500 cells/mm^3, *platelet count >/= 100,000 cells/mm^3, *Hgb >/= 9.0 g/dL.
* Patient has adequate liver function: *total bilirubin level </= 2.0 mg/dL, *albumin >/= 2.5 g/dL.
* Transaminases (SGOT and/or SGPT) may be up to 2.5 x ULN if alkaline phosphatase is </= ULN, or alkaline phosphatase may be up to 4 x ULN if transaminases are </= ULN.
* Patient has adequate renal function: a serum creatinine < 2 mg/dl
* Patient has signed a written informed consent.
* Patient has received no more than 2 prior chemotherapeutic regimens for recurrent or metastatic disease. Prior biologic therapy is not included.

Exclusion Criteria:

* Patient has received 3 or more prior chemotherapeutic regimens for recurrent/metastatic disease.
* No biopsy accessible tissue.
* Patient has received radiation therapy within the past 6 months.
* Prior radiation to the biopsy site.
* Patient has signs or symptoms of acute infection requiring systemic therapy.
* Patient exhibits confusion, disorientation, or has a history of major psychiatric illness which may impair patient's understanding of the informed consent.
* Patient has grade 3 or 4 neurotoxicity from previous anticancer treatment or significant neuropathy from any cause.
* Patient requires total parenteral nutrition with lipids.
* Surgery is anticipated to leave patient unable to swallow the SCH66336 or 4-HPR daily.
* Patient has a history of uncontrolled heart disease (including arrhythmia, angina, congestive heart failure, or any heart condition that cannot be controlled with regular ongoing medication)
* Because of the known teratogenic effect of retinoids, pregnant women and women who are currently breast-feeding may not participate in this study. All women of childbearing potential must have a negative pregnancy test within 24 hours prior to enrolling in the study.
* Serious infection or other intercurrent illness requiring immediate therapy.
* Inability to swallow oral medications, or other medical or social factors interfering with compliance.
* Patients may not take high dose synthetic or natural Vitamin A derivatives (>10,000 IU per day). Patients may not be taking high-dose vitamin A within 30 days of study entry.
* Patients should not take any anti-oxidants such as Vitamin E or Vitamin C
* Patients with pre-existing retinopathy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2005-01-20 (Actual); Primary Completion 2006-01 (Actual); Study Completion 2006-11 (Actual)

PRIMARY OUTCOMES:
Maximum Tolerated Dose (MTD) | 21 day courses
  MTD derived from lack of dose limiting toxicities (DLT) in 4 differing dose levels.

CONTACTS AND LOCATIONS:
Overall Officials: Edward S Kim, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- UT MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: UT MD Anderson Cancer Center website — http://www.mdanderson.org